CLINICAL TRIAL: NCT01425177
Title: Effect of Saline Irrigation to Decrease Rate of Residual Common Bile Duct Stones
Acronym: SIDEROD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sang Hyub Lee, Assistant Professor of Internal Medicine, Seoul National University Bundang Hospital, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LSH 0909
Record Dates: First submitted 2011-08-26; First posted 2011-08-29 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Common Bile Duct Gallstones
Keywords: Retained CBD Stones; Recurrent CBD Stones
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Normal saline irrigation (Experimental)
  Interventions: Procedure: Normal Saline Irrigation

INTERVENTIONS:
Procedure: Normal Saline Irrigation — After removing CBD stones with the ERCP, 200ml of the normal saline solution was irrigated into the common bile duct.

SUMMARY:
In recent years, endoscopic sphincterotomy and stone extraction are standard procedures for the removal of bile duct stones.

After procedures, there are some complications such as stone recurrence, papillary stenosis, cholangitis and liver abscess. These recurrent symptomatic bile duct stones, despite increasing experience and success with the procedure, occur in 4% to 24% of patients.

Gallbladder stone, pneumobilia and many other various factors are known to be associated with CBD stone recurrence. Lithotripsy was also related to the development of recurrent stones. It is natural that small stone fragments left after lithotripsy may act as nidi for stone recurrence.

Small remaining stone could not be completely detected only using ERCP stone removal and remaining stone removal can reduce residual and recurrent stones. Saline irrigation was effective immediately after ERCP stone removal to remove remaining small stones.

Saline irrigation has many advantages such as easy to treatment during ERCP stone removal, almost no additional cost and rare side effect. This study The authors expect this study is a remarkable role of ERCP stone removal procedure.

DETAILED DESCRIPTION:
CBD stones are defined as the occurrence of stones in the bile ducts. CBD stone usually causes biliary pain and jaundice, whereas obstruction that develops gradually over several months may manifest initially as pruritus or jaundice alone.

Unlike stones in the gallbladder, CBD stones cause symptoms, tend to present as life-threatening complications such as cholangitis and acute pancreatitis. Given its propensity to result in these serious complications, choledocholithiasis warrants treatment in nearly all cases In 2010, guideline for the risk and treatment of choledocholithiasis was published. The most predictive variables seem to be cholangitis, a bilirubin level higher than 1.7 mg/dL, and a dilated CBD on US. The presence of 2 or more of these variables results in a high probability of a CBD stone. Advanced age (older than 55 years), elevation of a liver biochemical test result other than bilirubin, and pancreatitis are less robust predictors for choledocholithiasis.

There are various ways of non invasive imaging diagnosis of CBD stone. The sensitivity of transabdominal US and conventional computed tomography (CT) in the detection of biliary stones is variable, ranging from 20% to 80% and from 23% to 85%, respectively. MRCP had sensitivity 92-93%, specificity 97-98%. Although MRCP is most excellent in diagnosis, the sensitivity is reduced 33-71% at diagnosis of small stones(less than 5mm) An ERCP has traditionally been considered the evaluation of biliary-tract diseases. This modality is very sensitive (90%) and specific (98%) in detecting CBD stone. EUS for the diagnosis of CBD stone reports widely varying sensitivities of 71% to 100% and specificities of 67% to 100%. Some papers report that intraductal ultrasound(IDUS) is very sensitive(97-100%). However, this is expensive and requires the fully-experienced endoscopist, so, it is difficult to use that.

In recent years, endoscopic sphincterotomy and stone extraction are standard procedures for the removal of bile duct stones. After procedures, there are some complications such as stone recurrence, papillary stenosis, cholangitis and liver abscess. These recurrent symptomatic bile duct stones, despite increasing experience and success with the procedure, occur in 4% to 24% of patients.

Retained stone is defined as incomplete stone removal during ERCP, otherwise recurrent stone is defined as recurrence stone after complete stone removal. A criterion to distinguish between the two is stones rediscovery time after ERCP stone removal. Typically, bile duct stones found 6 months or more after endoscopic retrograde cholangiopancreatography (ERCP) generally are considered recurrent, as opposed to retained Gallbladder stone, pneumobilia and many other various factors are known to be associated with CBD stone recurrence. Lithotripsy was also related to the development of recurrent stones. It is natural that small stone fragments left after lithotripsy may act as nidi for stone recurrence.

For this reason, many studies that reduce the residual and recurrence CBD stones have been performed. Before procedures, MRCP, CT and EUS are performed to identify the exact location of stones. Many studies demonstrated that residual stone clearance with ENBD, EUS or IDUS immediately after ERCP stone removal are useful in reducing the recurrence.

However, cholangiogram with ENBD or using EUS after ERCP stone removal increases the duration of hospital stay, cost and the patient's discomfort. Until now, non-invasive, time reduced, cheap and simply way was unknown.

Recently, two different studies were published. Using IDUS could effectively find residual CBD stones that persisted after EST and balloon and basket extraction. Furthermore, normal saline irrigation of CBD after stone removal appeared useful in clearing residual small stones. These procedures could reduce the retained and recurrent stone Another study showed that additional IDUS to confirm complete stone clearance after ERCP with basket stone removal significantly decreases the early recurrence rate of common bile duct stones.

These studies demonstrated that small remaining stone could not be completely detected only using ERCP stone removal and remaining stone removal can reduce residual and recurrent stones. Saline irrigation was effective immediately after ERCP stone removal to remove remaining small stones .

However, prospective study that saline irrigation without EUS or IDUS can reduce recurrent CBD stones after ERCP stone removal does not yet. Saline irrigation has many advantages such as easy to treatment during ERCP stone removal, almost no additional cost and rare side effect. This study The authors expect this study is a remarkable role of ERCP stone removal procedure.

ELIGIBILITY:
Inclusion Criteria:

* The patients were treated with CBD stone removal during therapeutic ERCP after finding CBD stones with CT, ultrasound or MRCP.
* The patients were treated with CBD stone removal during diagnostic ERCP because of cholangitis or cholecystitis.

Exclusion Criteria:

* Hemodynamic instability
* Younger than 18
* Mental illness
* Received previous CBD stone removal
* Hemolytic anemia, IHD stone, parasites in hepatobiliary system
* Genetic, autoimmune, congenital biliary disorder
* Liver or biliary surgery except cholecystectomy
* Pancreatic cancer, cholangiocarcinoma, ampulla of vater cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Retained CBD stones | From 3 to 6 months after procedure
  * CT or USG
  * Symptomatic choledocholithiasis

SECONDARY OUTCOMES:
Recurrent CBD Stones | Over 6months after procedure
  * CT, USG
  * Symptomatic choledocholithiasis
Cholangitis | Over 6months after procedure
  - Fever, RUQ pain, Jaundice

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hyub Lee, M.D. Ph.D, Study Director — Department of Internal Medicine, Seoul National University Bundang Hospital; Sang Eon Jang, M.D., Principal Investigator — Department of Internal Medicine, Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seoungnam, Gyeonggi-do, South Korea

REFERENCES:
- [Background] ASGE Standards of Practice Committee; Maple JT, Ben-Menachem T, Anderson MA, Appalaneni V, Banerjee S, Cash BD, Fisher L, Harrison ME, Fanelli RD, Fukami N, Ikenberry SO, Jain R, Khan K, Krinsky ML, Strohmeyer L, Dominitz JA. The role of endoscopy in the evaluation of suspected choledocholithiasis. Gastrointest Endosc. 2010 Jan;71(1):1-9. doi: 10.1016/j.gie.2009.09.041. No abstract available. PMID 20105473
- [Background] Einstein DM, Lapin SA, Ralls PW, Halls JM. The insensitivity of sonography in the detection of choledocholithiasis. AJR Am J Roentgenol. 1984 Apr;142(4):725-8. doi: 10.2214/ajr.142.4.725. PMID 6608231
- [Background] Miller FH, Hwang CM, Gabriel H, Goodhartz LA, Omar AJ, Parsons WG 3rd. Contrast-enhanced helical CT of choledocholithiasis. AJR Am J Roentgenol. 2003 Jul;181(1):125-30. doi: 10.2214/ajr.181.1.1810125. No abstract available. PMID 12818842
- [Background] Soto JA, Alvarez O, Munera F, Velez SM, Valencia J, Ramirez N. Diagnosing bile duct stones: comparison of unenhanced helical CT, oral contrast-enhanced CT cholangiography, and MR cholangiography. AJR Am J Roentgenol. 2000 Oct;175(4):1127-34. doi: 10.2214/ajr.175.4.1751127. PMID 11000177
- [Background] Boraschi P, Neri E, Braccini G, Gigoni R, Caramella D, Perri G, Bartolozzi C. Choledocolithiasis: diagnostic accuracy of MR cholangiopancreatography. Three-year experience. Magn Reson Imaging. 1999 Nov;17(9):1245-53. doi: 10.1016/s0730-725x(99)00075-2. PMID 10576709
- [Background] Tse F, Liu L, Barkun AN, Armstrong D, Moayyedi P. EUS: a meta-analysis of test performance in suspected choledocholithiasis. Gastrointest Endosc. 2008 Feb;67(2):235-44. doi: 10.1016/j.gie.2007.09.047. PMID 18226685
- [Background] Das A, Isenberg G, Wong RC, Sivak MV Jr, Chak A. Wire-guided intraductal US: an adjunct to ERCP in the management of bile duct stones. Gastrointest Endosc. 2001 Jul;54(1):31-6. doi: 10.1067/mge.2001.115006. PMID 11427838
- [Background] Tseng LJ, Jao YT, Mo LR, Lin RC. Over-the-wire US catheter probe as an adjunct to ERCP in the detection of choledocholithiasis. Gastrointest Endosc. 2001 Dec;54(6):720-3. doi: 10.1067/mge.2001.119255. PMID 11726847
- [Background] Cotton PB, Geenen JE, Sherman S, Cunningham JT, Howell DA, Carr-Locke DL, Nickl NJ, Hawes RH, Lehman GA, Ferrari A, Slivka A, Lichtenstein DR, Baillie J, Jowell PS, Lail LM, Evangelou H, Bosco JJ, Hanson BL, Hoffman BJ, Rahaman SM, Male R. Endoscopic sphincterotomy for stones by experts is safe, even in younger patients with normal ducts. Ann Surg. 1998 Feb;227(2):201-4. doi: 10.1097/00000658-199802000-00008. PMID 9488517
- [Background] Duensing RA, Williams RA, Collins JC, Wilson SE. Managing choledocholithiasis in the laparoscopic era. Am J Surg. 1995 Dec;170(6):619-23. doi: 10.1016/s0002-9610(99)80028-2. PMID 7492013
- [Background] Keizman D, Shalom MI, Konikoff FM. An angulated common bile duct predisposes to recurrent symptomatic bile duct stones after endoscopic stone extraction. Surg Endosc. 2006 Oct;20(10):1594-9. doi: 10.1007/s00464-005-0656-x. Epub 2006 Jul 20. PMID 16858527
- [Background] Cheon YK, Lehman GA. Identification of risk factors for stone recurrence after endoscopic treatment of bile duct stones. Eur J Gastroenterol Hepatol. 2006 May;18(5):461-4. doi: 10.1097/00042737-200605000-00001. PMID 16607138
- [Background] Ando T, Tsuyuguchi T, Okugawa T, Saito M, Ishihara T, Yamaguchi T, Saisho H. Risk factors for recurrent bile duct stones after endoscopic papillotomy. Gut. 2003 Jan;52(1):116-21. doi: 10.1136/gut.52.1.116. PMID 12477771
- [Background] Tsuchiya S, Tsuyuguchi T, Sakai Y, Sugiyama H, Miyagawa K, Fukuda Y, Ando T, Saisho H, Yokosuka O. Clinical utility of intraductal US to decrease early recurrence rate of common bile duct stones after endoscopic papillotomy. J Gastroenterol Hepatol. 2008 Oct;23(10):1590-5. doi: 10.1111/j.1440-1746.2008.05458.x. Epub 2008 Jun 12. PMID 18554235
- [Background] Ang TL, Teo EK, Fock KM, Lyn Tan JY. Are there roles for intraductal US and saline solution irrigation in ensuring complete clearance of common bile duct stones? Gastrointest Endosc. 2009 Jun;69(7):1276-81. doi: 10.1016/j.gie.2008.10.018. Epub 2009 Feb 26. PMID 19249039
- [Background] Boix J, Lorenzo-Zuniga V, Ananos F, Domenech E, Morillas RM, Gassull MA. Impact of periampullary duodenal diverticula at endoscopic retrograde cholangiopancreatography: a proposed classification of periampullary duodenal diverticula. Surg Laparosc Endosc Percutan Tech. 2006 Aug;16(4):208-11. doi: 10.1097/00129689-200608000-00002. PMID 16921297
- [Derived] Ahn DW, Lee SH, Paik WH, Song BJ, Park JM, Kim J, Jeong JB, Hwang JH, Ryu JK, Kim YT. Effects of Saline Irrigation of the Bile Duct to Reduce the Rate of Residual Common Bile Duct Stones: A Multicenter, Prospective, Randomized Study. Am J Gastroenterol. 2018 Apr;113(4):548-555. doi: 10.1038/ajg.2018.21. Epub 2018 Mar 27. PMID 29610513
- See also: Seoul National University Bundang Hospital — http://www.snubh.org/
- See also: Seoul National University College of Medicine — http://medicine.snu.ac.kr/
- See also: Korea Food and Drug Administration — http://www.kfda.go.kr/